CLINICAL TRIAL: NCT02331537
Title: Internet-based Exposure Therapy for Excessive Worry: A Randomized Trial
Brief Title: Internet-based Exposure Therapy for Excessive Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1944-31-5
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Excessive Worry; Rumination
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based cognitive-behavior therapy (Experimental): The experimental group will go through active internet-based treatment. The treatment is 10 weeks long and is based on the principles of exposure i.e. the participant is instructed to stay with the frightening thought until it is no longer associated with anxiety.
  Interventions: Behavioral: Internet-based cognitive-behavior therapy
- Waitlist (No Intervention): Waitlist control that will get the internet-based treatment when the first group has finished (i.e. Week 10). There are no active treatment for these participants at all.

INTERVENTIONS:
Behavioral: Internet-based cognitive-behavior therapy — Internet-based cognitive-behavior therapy on a safe internet platform. Treatment is divided into seven modules, each containing homework assignments . The participants will be assigned a therapist that they can contact through a message system in the platform and expect answer within 24 hours.
  Arms: Internet-based cognitive-behavior therapy

SUMMARY:
The purpose of this study is to examine if an internet-based exposure therapy is effective in reducing excessive worry amongst patients who suffer from this problem.

DETAILED DESCRIPTION:
Trial Objectives: Primary objective is to investigate whether an Internet-based exposure therapy can effectively reduce the degree of excessive worry. The secondary objective is to a) investigate whether imagery based exposure is more effective than verbal exposure. b) investigate the cost-effectiveness of this treatment and c) to study if any variables could moderate/mediate the treatment outcome, such as metacognitions, degree of rumination or degree of depression.

Trial Design: Randomized controlled trial with waitlist control, who also will recieve treatment after the first group has finished.

Duration: Ten weeks

Primary Endpoint: Change in worry symptoms from baseline to Week 10. Long term follow-up is also investigated (baseline to 4-months after treatment completion and baseline to 12-months after treatment completion).

Efficacy Parameters: Penn State Worry Questionnaire (PSWQ)

Safety Parameters: Adverse Events is assessed weekly via the internet.

Description of Trial Subjects: Patients > 18 years old with a PSWQ score more than 56 points

Number of Subjects: 140

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* ≥ 18 years
* Situated in Sweden
* Informed consent
* Penn State Worry Questionnaire score more than 56 points

Exclusion Criteria:

* Substance dependence during the last six months
* Post traumatic stress disorder, bipolar disorder or psychosis
* Symptoms better explained by axis 2 diagnosis (e.g. autism or borderline personality disorder)
* MADRS-S score above 25 points
* Psychotropic medication changes within two months prior to treatment that could affect target symptoms.
* Received exposure based Cognitive behavior therapy (CBT) for pathological worry the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Week 0, Week 10, Long term follow-up at 4-, and 12-months after treatment has ended
  Change in worry from baseline to Week 10, and at 4- and 12 months after treatment has ended.

SECONDARY OUTCOMES:
Meta Cognitions Questionnaire (MCQ-30) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in metacognitions from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in depression from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Euroqol (EQ-5D) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in general health from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Hospital anxiety and depression scale (HADS) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in anxiety and depression from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Spontaneous Use of Imagery Scale (SUIS) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in Spontaneous Use of Imagery from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Cognitive Avoidance Questionnaire (CAQ) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in cognitive avoidance from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in economic costs from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Intolerance of Uncertainty Scale (IUS) | Week 0, Week 10, long term follow-up at 4- and 12- months after treatment has ended
  Change in tolerance of uncertainty from baseline to Week 10 and at 4- and 12 months after treatment has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden